CLINICAL TRIAL: NCT03832777
Title: Effect of Transcranial Magnetic Stimulation on Dorsomedial Cortex in Clinical and Neuropsychological Variables in Borderline Personality Disorder
Brief Title: Transcranial Magnetic Stimulation on Dorsomedial Prefrontal Cortex in Borderline Personality Disorder
Acronym: TMS&BPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de Queretaro (Other)
Responsible Party: Principal Investigator, Dr. Julian Reyes López, Professor, Universidad Autonoma de Queretaro
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 04-01/02/2018
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Personality Disorders
MeSH Terms: conditions — Borderline Personality Disorder; Personality Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The aim of this study is to evaluate the clinical effects of 5Hz rTMS over Dorsomedial Prefrontal Cortex on an active versus placebo modality stimulation.
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 Hz Stimulation (Active Comparator): This group will receive 5Hz (Hertz) Dorsomedial Prefrontal Cortex repetitive Transcranial Magnetic Stimulation with 1500 pulses per session, once per weekday, with a final result of 15 sessions in this modality.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Placebo Stimulation (Placebo Comparator): This group will receive the Sham modality simulating 1500 pulses of 5Hz Transcranial Magnetic Stimulation for 15 sessions, one per weekday.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Subjects will receive both active and placebo rTMS, in a crossover modality.
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
This study evaluates the effect of 5Hz repetitive Transcranial Magnetic Stimulation (rTMS) on Dorsomedial Prefrontal Cortex on Borderline Personality Disorder (BPD).

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is a mental illness with a high worldwide prevalence and economic costs, and is characterized with impulsiveness, both interpersonal relationships and emotional disturbance. Symptoms are related to hypofunction of frontal areas like Dorsomedial Prefrontal Cortex (DMPFC). Psychotherapy is the base treatment in this disease, but economic costs and long-time therapy have made difficult the attachment. Repetitive Transcranial Magnetic Stimulation(rTMS), authorized by Food and Drug Administration (FDA) on Major Depressive Disorder (MDD) treatment has proven good results in previous works in BPD clinical characteristics on both dorsolateral prefrontal cortex (DLPFC) and enhancement in depressive symptoms stimulating DMPFC in high frequency. However, there are no current research that have addressed the use of low-frequency on this anatomical area.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old.
* Meet DSM 5 (Diagnostic and Statistical Manual, 5th edition) diagnostic criteria for Borderline Personality Disorder.
* Score of >7 in the Diagnostic Interview for Borderline (Revised version, DIB-R)
* All patients must have follow-up psychotherapy of at least one month.
* No changes on pharmacological treatment within the last month.
* Patients must provide their oral and written informed consent.

Exclusion Criteria:

* Subjects with history of traumatic brain injury with loss of consciousness.
* Subjects with intracranial metallic objects or metal plates in the skull.
* Subjects diagnosed with uncontrolled chronic (for example: hypertension, diabetes) or neurological diseases.
* Comorbidity with other mental illness. (Except Depressive symptoms and Anxiety Disorders).
* Presence of psychotic symptoms.
* Alterations in the electroencephalogram (epileptiform activity).
* Self injury or suicidal attempts in less than 2 weeks (depends on the severity and deepness).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Borderline Symptoms List (BSL) | 6 weeks
  BSL is a 23 item scale that evaluates the general symptoms and 11 items with behavioural evaluation of BPD.
Global Clinical Impression of BPD (GCI-BPD) | 6 weeks
  CGI-BPD is a 10 item evaluation that rates the severity of BPD distributed in 9 neuropsychological domains with a final global score.
Borderline Evaluation of Severity Over Time (BEST) | 6 weeks
  BEST is a 15 item scale that evaluates the severity in this pathology according to 3 areas: thoughts, emotions and typical behaviours.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | 6 weeks
  HDRS is a 21 item scale that evaluates the severity of depressive symptoms in patients.
Hamilton Anxiety Rating Scale (HARS) | 6 weeks
  HARS is a 14 items rating scale that evaluates the severity of anxiety symptoms in patients.
Barratt Impulsivity Scale (BIS-11) | 6 weeks
  The Barratt Impulsiveness Scale is a questionnaire designed to assess the personality / behavioral construct of impulsiveness; composed of 30 items describing common impulsive or non-impulsive (for reversed scored items) behaviors and preferences .

CONTACTS AND LOCATIONS:
Overall Officials: Julian V Reyes-López, Psychiatrist, Study Director — Faculty of Medicine, Autonomous University of Queretaro
Locations (1):
- Autonomous University of Queretaro, Querétaro City, Querétaro, Mexico

REFERENCES:
- [Derived] Calderon-Moctezuma AR, Reyes-Lopez JV, Rodriguez-Valdes R, Barbosa-Luna M, Ricardo-Garcell J, Espino-Cortes M, Hernandez-Chan N, Garcia-Noguez L, Roque-Roque G, Trejo-Cruz G, Canizares-Gomez S, Hernandez-Montiel H. Improvement in borderline personality disorder symptomatology after repetitive transcranial magnetic stimulation of the dorsomedial prefrontal cortex: preliminary results. Braz J Psychiatry. 2021 Feb 1;43(1):65-69. doi: 10.1590/1516-4446-2019-0591. eCollection 2020. PMID 32876128